CLINICAL TRIAL: NCT05805410
Title: Neuromuscular Mechanisms of Specific Trunk Interventions in Children With Cerebral Palsy
Brief Title: Neuromuscular Mechanisms of Specific Trunk Interventions in Children With CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Ming Wu, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS115487 (NIH)
Record Dates: First submitted 2022-12-07; First posted 2023-04-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic hippotherapy (Experimental): For the robotic training group, each subject will be trained for 40 minutes. Specifically, each participant will sit astride on a robotic horse with the force perturbation will be applied in the anterior-posterior direction and up/down direction.
  Interventions: Behavioral: robotic hippotherapy
- Conventional physical therapy (Active Comparator): For the conventional physical therapy group, each subject will be trained for 40 minutes, which will include 10 minutes of stretching, followed by 10 minutes of sitting and 10 minutes of standing balance training, and 10 minutes of treadmill walking.
  Interventions: Behavioral: Conventional physical therapy

INTERVENTIONS:
Behavioral: robotic hippotherapy — A custom designed cable-driven robotic system that mimics horseback movement during walking was used in this study.
  Arms: Robotic hippotherapy
Behavioral: Conventional physical therapy — Stretching of trunk and leg muscles, followed by sitting and standing balance training, and conventional treadmill walking.
  Arms: Conventional physical therapy

SUMMARY:
Determine the effect of repeated pelvis perturbation training on trunk posture and locomotor function in children with CP.

DETAILED DESCRIPTION:
We will determine whether repeat exposure to pelvis perturbation during sitting astride will induce functional improvements in trunk postural control and locomotion in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of bilateral spastic CP attributed to complications of prematurity, intracranial hemorrhage and periventricular leukmalacia according to the definition of Bax.
* Children aged 4 to 12 years old without Botulinum toxin treatment within 6 months, and without surgeries (such as selective dorsal rhizotomy) within 12 months before the onset of the training.
* Subjects will be able to remain seated without help for ≥10s.
* GMFCS levels will be I to IV.
* Children must be able to signal pain, fear or discomfort reliably.
* Children with mild scoliosis (Cobb angle < 20 °).
* Children with CP who have no prior hippotherapy experiences within 6 months.

Exclusion Criteria:

* severe lower extremity contractures, fractures, osseous instabilities, osteoporosis.
* severe disproportional bone growth.
* unhealed skin lesions in the lower extremities.
* thromboembolic diseases, cardiovascular instability.
* aggressive or self-harming behaviors.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Trunk Control Measurement Scale (TCMS) score from baseline. | baseline, post 6 weeks of training and 8 weeks after the end of training.
  The maximum value for the total TCMS is 58 points (no unit). Specifically, there is 20 points for the category 'static sitting balance', 28 points for 'selective movement control', and 10 points for 'dynamic reaching'). A higher TCMS scores indicates a better motor performance in trunk control.

SECONDARY OUTCOMES:
Change in Walking speed from baseline | baseline, post 6 weeks of training and 8 weeks after the end of training.
  Overground walking speed
Chang in 6-minute walking distance from baseline | baseline, post 6 weeks of training and 8 weeks after the end of training.
  Walking distance within 6 minutes
Change in GMFM-66 | baseline, post 6 weeks of training and 8 weeks after the end of training.
  Gross Motor Function Measure

CONTACTS AND LOCATIONS:
Overall Officials: Ming Wu, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No